CLINICAL TRIAL: NCT00013338
Title: Supported Treadmill Ambulation Training After Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: B2142R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury, ambulation, treadmill
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Ambulation Training

SUMMARY:
This is a randomized, controlled trial to compare supported treadmill ambulation training (STAT) to conventional gait training for improving gait speed, gait endurance, gait efficiency and muscle function in SCI subjects injured more than six months prior to start of training. Each subject will receive twelve weeks of either CGT or STAT, given as 20 minutes of training within a one-hour period per day, five days per week. These subjects will be studied baseline, 4,8 and 12 weeks of training, and three months after the end of training with a battery of tests designed to evaluate the subjects' gait and muscle function.

ELIGIBILITY:
Spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2000-01; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Program Analysis and Review Section (PARS), Department of Veterans Affairs, Rehabilitation Research and Development Service; Nancy Rocheleau, Program Analyst — Program Analysis and Review Section (PARS), Department of Veterans Affairs, Rehabilitation Research and Development Service
Locations (1):
- VAMC, Houston, Houston, Texas, United States